CLINICAL TRIAL: NCT01754987
Title: Phase I/II Study of Intravenous Ascorbic Acid in Treatment of Metastatic Hepatocellular Carcinoma
Brief Title: A Study of Vitamin C in the Treatment of Liver Cancer to Determine if it is Safe and Effective
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12D.424; JT 2306 (Other: JeffTrial Number)
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Hepatocellular Carcinoma; Advanced Liver Cancer
Keywords: Vitamins; Malignant Tumor, Tumour; Integrative Medicine; Complementary Medicine; Alternative Medicine Antioxidants; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Protective Agents; Physiological Effects of Drugs; Micronutrients; Growth Substances; Antineoplastic Agents, Phytogenic; Antineoplastic Agents; Therapeutic Uses; Radiation-Sensitizing Agents; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Liver Neoplasms | interventions — Ascorbic Acid; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ascorbic Acid + Sorafenib (Experimental): Drug: Vitamin C Other Names: Ascorbic Acid, Ascorbate
  Dosage:
  Vitamin C : 100 grams (infusion) Phase I: 3x a week for 8 weeks Phase II: 3x a week for 16 weeks Sorafenib: taken daily (oral)
  Interventions: Drug: Ascorbic Acid + Sorafenib
- Sorafenib alone (Other): Sorafenib: taken daily (oral)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Ascorbic Acid + Sorafenib
  Other Names: Vitamin C; Ascorbate
  Arms: Ascorbic Acid + Sorafenib
Drug: Sorafenib
  Other Names: Nexavar
  Arms: Sorafenib alone

SUMMARY:
This protocol is a phase I/II, study of ascorbic acid (AA) infusions combined with treatment with sorafenib versus treatment with sorafenib alone in subjects with metastatic hepatocellular carcinoma. The phase I aspect will assess the safety and efficacy of the concurrent treatments and the phase II aspect will utilize CT (computer-tomography) scans to assess overall tumor response rate and evaluate disease progression

DETAILED DESCRIPTION:
Intravenous Ascorbic Acid (Vitamin C) is a widely used alternative cancer treatment. This trial will study an intravenous Vitamin C treatment for persons with liver cancer that has spread, who are also receiving Sorafenib (a standard cancer drug), to see whether the combination of Vitamin C and Sorafenib is safe and well tolerated. Phase I will involve 6 persons who will receive the Vitamin C for 8 weeks to more specifically assess the safety of getting Vitamin C in combination with Sorafenib. Phase II will be randomized to receive either Vitamin C plus Sorafenib or Sorafenib alone for 16 weeks. If Vitamin C has a beneficial effect on tumour cells, patients may experience a regression of tumor or tumor markers. Additional benefits include scans at no charge to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Metastatic hepatocellular carcinoma
* G6PD (glucose-6-phosphate dehydrogenase) status > lower limit of normal
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Laboratory at baseline evaluation for inclusion in the study: creatinine ≤1.5X upper limit (if the creatinine is elevated, but ≤1.5X the ULN, a 24 hour creatinine clearance will be obtained); transaminase (AST/ALT) ≤2.0X upper limit of normal; bilirubin levels ≥ 2 mg/dL; ANC ≥1,500/mm3; Hemoglobin > 8g/dL; platelet ≥ 100,000/mm3
* Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the study.
* Willing and able to provide informed consent and participate in the study procedures.

Exclusion Criteria:

* Patients with evidence of a significant current psychiatric disorder that would prevent completion of the study as determined by the PI will not be allowed to participate.
* Co-morbid medical condition that would affect survival or tolerance as determined by the PI. This includes patients who have not fully recovered from toxicities associated with prior therapy. It also includes subjects who, as determined by the PI, are at risk of experiencing fluid overload (i.e., congestive heart failure).
* Patients who currently abuse alcohol or drugs.
* Patients with known glomerular filtration rate of <60ml/min or with nephrotic range proteinuria.
* Pregnant or lactating women
* Enrollment in active clinical trial/ experimental therapy or IND study within the prior 30 days.
* Contraindication for CT or PET/CT as per the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Monti, MD, MBA, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monti DA, Mitchell E, Bazzan AJ, Littman S, Zabrecky G, Yeo CJ, Pillai MV, Newberg AB, Deshmukh S, Levine M. Phase I evaluation of intravenous ascorbic acid in combination with gemcitabine and erlotinib in patients with metastatic pancreatic cancer. PLoS One. 2012;7(1):e29794. doi: 10.1371/journal.pone.0029794. Epub 2012 Jan 17. PMID 22272248

RESULTS

PARTICIPANT FLOW:
Groups:
- Ascorbic Acid + Sorafenib: Drug: Vitamin C Other Names: Ascorbic Acid, Ascorbate
  Dosage:
  Vitamin C : 100 grams (infusion) Phase I: 3x a week for 8 weeks Phase II: 3x a week for 16 weeks Sorafenib: taken daily (oral)
  Ascorbic Acid + Sorafenib
- Sorafenib Alone: Sorafenib: taken daily (oral)
  Sorafenib
Period: Overall Study
Arm/Group | Ascorbic Acid + Sorafenib | Sorafenib Alone
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The trial was terminated prematurely. No patients were accrued to the Sorafenib arm. Data were not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Ascorbic Acid + Sorafenib | Sorafenib Alone | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 2 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 5 |  | 5
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience Serious Adverse Events.
Description: The primary aim is to assess whether or not (IV) Ascorbic Acid (AA) with sorafenib therapy is relatively safe and well-tolerated according to Common Terminology Criteria for Adverse Events (CTCAE)v4.0
Time Frame: 16 weeks +/- 2 weeks
Population: The trial was closed early due to lack of accrual. The data were not collected or analyzed.
Arm/Group | Ascorbic Acid + Sorafenib | Sorafenib Alone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Tumor Response Rate
Description: To utilize CT or PET/CT scans to assess overall tumor response rate (complete) in subjects with advanced metastatic hepatocellular cancer treated with the combination of ascorbic acid and sorafenib versus sorafenib alone.
Time Frame: 16 weeks +/- 2 weeks
Population: The trial was closed early due to lack of accrual. The data were not collected or analyzed.
Arm/Group | Ascorbic Acid + Sorafenib | Sorafenib Alone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Value Collected Using the Functional Assessment of Cancer Therapy-General (FACT-G) Quality Assessment Instrument
Description: To evaluate quality of life using Functional Assessment of Cancer Therapy-General (FACT-G) quality assessment instrument. The FACT-G questionnaire will be used to assess quality-of-life longitudinally. Quality-of-life scores obtained from the FACT-G will be summarized at multiple time points. Five-point scale from 0 (not at all) to 4 (very much)
Time Frame: 16 weeks +/- 2 weeks
Population: The trial was closed early due to lack of accrual. The data were not collected or analyzed.
Arm/Group | Ascorbic Acid + Sorafenib | Sorafenib Alone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants That Are Alive After 15 Weeks of Treatment.
Description: To evaluate duration of tumor response and progression-free survival
Time Frame: 15 weeks+
Population: The trial was closed early due to lack of accrual. The data were not collected or analyzed.
Arm/Group | Ascorbic Acid + Sorafenib | Sorafenib Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ascorbic Acid + Sorafenib | Sorafenib Alone
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 2/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid + Sorafenib (N=5) | Sorafenib Alone (N=0)
Dehydration (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbic Acid + Sorafenib (N=5) | Sorafenib Alone (N=0)
Elevated Creatinine (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Nosebleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low Platelet count (Blood and lymphatic system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes